CLINICAL TRIAL: NCT06506448
Title: Anatomical, Physiological and Inflammatory Characterization of the Non-Culprit Vessels in Patients Undergoing Primary PCI for ST-Elevation Myocardial Infarction in the Presence of Multivessel Disease Toward a Personalised Approach to Complete Revascularisation After Primary PCI
Brief Title: Risk Characterization of Non-culprit Vessels in Patients Undergoing Primary PCI for ST-elevation MI in Multivessel Disease
Acronym: PICNIC
Status: Recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Boston Scientific Corporation (Industry); HeartFlow, Inc. (Industry); Wessex Heartbeat (Unknown); Caristo (Unknown)
Responsible Party: Sponsor
Other Study IDs: RHMCAR0647
Record Dates: First submitted 2024-05-22; First posted 2024-07-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Primary percutaneous coronary intervention; Infarct related artery; Non-infarct related artery; Computerised Tomography Coronary Angiography CTCA; Fractional Flow Reserve from CT (FFRct); Fat Attenuation Index (FAI); Inflammation
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Single blood sample taken from participants at baseline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- STEMI patients with multivessel disease: 320 patients undergoing primary angioplasty for ST-elevation myocardial infarction (STEMI) who have bystander disease in a main coronary artery with at least one stenosis of 50% or more
  Interventions: Diagnostic Test: CT Coronary Angiography

INTERVENTIONS:
Diagnostic Test: CT Coronary Angiography — CTCA for anatomical, physiological, plaque composition and inflammatory assessment of coronary arteries
  Other Names: FFRCT and plaque analysis (HeartFlow) and Fat Attenuation Index (Caristo)

SUMMARY:
Most heart attacks occur because a clot forms in a coronary artery blocking blood flow. Without blood heart muscle dies. Untreated, clots can cause a specific type of heart attack -ST-elevation myocardial infarction (STEMI). STEMI patients are treated immediately by finding the blocked artery ("culprit" lesion) using a dye injected into the coronary arteries and then by unblocking the artery using balloons and stents. This procedure - primary angioplasty - is offered 24/7 and limits the size of heart attacks and saves lives.

Cardiologists know how to treat STEMI patients but it's less clear what to do about narrowings in other coronary arteries ("bystander" disease). This is important - if they're left alone some bystander lesions can cause future events including heart attacks or angina. Recent trials compared stenting ALL the bystander narrowings after primary angioplasty, with stenting none and showed some benefit from stenting all of them ("complete revascularisation").

However, complete revascularisation carries extra risk, putting patients through more complicated procedures and using up resource. A blanket strategy of complete revascularisation of ALL bystander narrowings in ALL STEMI patients is unlikely to be the correct answer as only a small minority of these patients have further events.

In PICNIC the investigators want to identify bystander narrowings most likely to cause a future event, and those unlikely to do so. The study can then test the hypothesis that only the high-risk bystander narrowings need stenting, and the others can be treated with tablets only. Investigators will study patients using specialised imaging techniques from coronary artery CT scans and levels of inflammation to see which narrowings cause future events and which do not. If this can be done, a case can be made to test complete revascularisation only in bystander narrowings that look high risk.

DETAILED DESCRIPTION:
Approximately 50% of patients presenting with an acute ST-segment elevation myocardial infarction (STEMI) have multivessel coronary artery disease (CAD). Five randomized studies have shown that complete revascularization, either at the time of primary percutaneous coronary intervention (PPCI) or within 45 days of the index admission, is safe and reduces the risk of repeat coronary revascularization and myocardial infarction (MI), particularly in the non-infarct related artery (NIRA). Despite these improvements in clinical outcomes, no study to date has provided a mechanistic insight as to how complete revascularization of chronic bystander disease may lead to the observed benefit. Indeed, the randomized studies, through the variable nature of their results (reduction in MI versus revascularization etc), have suggested the possibility that there are differing mechanisms for the observed benefit. The data would also be consistent with the concept that not all patients undergoing primary PCI with bystander disease require or benefit from complete revascularisation. This is an important possibility with important potential implications for resource utilisation and patient experience.

The investigators hypothesize that the susceptibility of non-culprit disease to ischaemic events after primary PCI is variable between individuals, and possibly even between their coronary vessels and lesions. Specifically, the investigators postulate that this susceptibility may be related to multiple factors including their anatomical and physiological vulnerability, and their local vascular inflammatory status. In order to test this hypothesis, the investigators will systematically examine the following parameters in each bystander coronary vessel in patients who present with STEMI and are undergoing primary PCI of the culprit vessel:

1. markers of systemic inflammatory status
2. plaque anatomy including lesion severity and markers of lesion vulnerability on CTCA
3. assessment of individual coronary vessel inflammation using CT-derived fat attenuation index
4. vessel physiology using FFRCT (fractional flow reserve from computed tomography) incorporating wall shear stress and axial plaque stress.

Aims

The aims of this study are to address the following research questions:

1. What are the anatomical, physiological & inflammatory features of lesions in the NIRA(s) of patients presenting with STEMI who are treated with a strategy of culprit-only PPCI?
2. Is there an association between these anatomical, physiological & inflammatory features and the risk of non-culprit lesions causing adverse events in STEMI patients with significant bystander disease in the NIRA(s)?

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent (post PPCI)
2. Age 18 years to 85 years
3. Presentation of acute STEMI within 12 hours of symptom on-set
4. Culprit artery PPCI
5. Coronary stenosis of > 50% diameter stenosis by visual estimation in NIRA with a minimum diameter of 2.5mm

Exclusion Criteria:

1. Cardiogenic shock
2. Decompensated heart failure requiring intubation, inotropes, or intra-aortic balloon counter pulsation
3. Refractory ventricular arrhythmia
4. Previous coronary artery bypass surgery (CABG)
5. Stent thrombosis and in stent restenosis
6. An intention before inclusion into the study to revascularize a non-culprit lesion
7. Active malignancy or inflammatory disorders such as rheumatoid arthritis or inflammatory bowel disease
8. Severe valvular heart disease requiring surgery
9. Planned surgical revascularisation
10. Active participation in another study/trial
11. < 12 months life expectancy
12. Contraindication to CTCA

    * Presence of internal defibrillator
    * Known allergy to iodinated contrast
    * Pregnancy
    * Contraindication to intravenous beta blockade
    * Contraindication to acute sublingual nitrate administration
    * Mechanical prosthetic heart valve
    * Advanced renal impairment (creatinine >200)
    * Significant valve disease (sever aortic stenosis or regurgitation; severe mitral regurgitation)

Angiographic exclusion criteria

1. NIRA stenosis of 50% or more in the left main stem or the ostia of both the left anterior descending and circumflex arteries
2. < TIMI (thrombolysis in myocardial infarction) flow grade 3 in the NIRA,
3. Evidence of thrombus in the NIRA.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with ST elevation myocardial infarction who are found to have significant stenoses in the non-infarct related artery(s) defined as coronary stenosis >50% by visual estimation
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between major adverse cardiac & cerebrovascular events (MACCE) and CTCA-derived anatomical, physiological, plaque & inflammatory characteristics and serum inflammatory markers at 2 years | 2 years
  Correlation between:
  1. major adverse cardiac & cerebrovascular events (MACCE) defined as the composite of all-cause mortality, cardiovascular death, cardiac arrest, acute coronary syndrome (unstable angina, NSTEMI, or STEMI), additional revascularization by CABG or PCI, rehospitalisation for angina, heart failure, stroke, ventricular or atrial fibrillation or tachyarrhythmia at 2 years &:
  2. Anatomical & physiological characteristics of coronary vessels/lesions in the NIRA(s) as assessed by CTCA parameters (FFRCT + FAI + plaque characteristics)

SECONDARY OUTCOMES:
Correlation between major adverse cardiac & cerebrovascular events (MACCE) and components of CTCA-derived anatomical, physiological, plaque & inflammatory characteristics and serum inflammatory markers at 1 year | 1 year
  Correlation between:
  1. major adverse cardiac & cerebrovascular events (MACCE) defined as the composite of all-cause mortality, cardiovascular death, cardiac arrest, acute coronary syndrome (unstable angina, NSTEMI, or STEMI), additional revascularization by CABG or PCI, rehospitalisation for angina, heart failure, stroke, ventricular or atrial fibrillation or tachyarrhythmia at 1 year &:
  2. Anatomical & physiological characteristics of coronary vessels/lesions in the NIRA(s) as assessed by CTCA/FFRCT/FAI parameters between individual components of MACCE
Correlation between anatomical, physiological & serum inflammatory markers and future adverse events at 3 years | 3 years
  Correlation between:
  1. major adverse cardiac & cerebrovascular events (MACCE) defined as the composite of all-cause mortality, cardiovascular death, cardiac arrest, acute coronary syndrome (unstable angina, NSTEMI, or STEMI), additional revascularization by CABG or PCI, rehospitalisation for angina, heart failure, stroke, ventricular or atrial fibrillation or tachyarrhythmia at 3 years &:
  2. Anatomical & physiological characteristics of coronary vessels/lesions in the NIRA(s) as assessed by CTCA/FFRCT/FAI parameters between individual components of MACCE
Development of a risk score to predict clinical events based upon individual-, vessel- & lesion-specific factors | 1 year
  To build a multidimensional AI-mediated deep learning model that uses the following data inputs (a) blood biomarkers, (b) CTCA lesion severity, (c) CTCA conventional plaque characteristics (e.g. spotty calcification etc); (d) FFRCT-derived plaque characteristic (ie adverse plaque and haemodynamic characteristics); (d) FAI-derived output; (e) clinical characteristics in order to correlate them with clinical events. The model will then be used to develop a risk score
Development of a risk score to predict clinical events based upon individual-, vessel- & lesion-specific factors | 3 years
  To build a multidimensional AI-mediated deep learning model that uses the following data inputs (a) blood biomarkers, (b) CTCA lesion severity, (c) CTCA conventional plaque characteristics (e.g. spotty calcification etc); (d) FFRCT-derived plaque characteristic (ie adverse plaque and haemodynamic characteristics); (d) FAI-derived output; (e) clinical characteristics in order to correlate them with clinical events. The model will then be used to develop a risk score

CONTACTS AND LOCATIONS:
Overall Officials: Nick Curzen, PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - University Hospitals Dorset NHS Foundation Trust, Bournemouth, Dorset
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire

IPD SHARING:
Plan to Share IPD: No
Not applicable. There will be no individual participant data available to other researchers.